CLINICAL TRIAL: NCT05267925
Title: Single-arm, Open Label Clinical Trial of CuraLin in Type 2 Diabetes
Brief Title: CuraLin Herbal Supplement for Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending additional product QA
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBKK8321
Record Dates: First submitted 2022-01-03; First posted 2022-03-07 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will be asked to take the dietary herbal supplement CuraLin for the duration of the study. All participants will take 2 capsules orally, three times per day following meals for 12 weeks.
  Interventions: Dietary Supplement: CuraLin

INTERVENTIONS:
Dietary Supplement: CuraLin — CuraLin™ is a dietary supplement manufactured by NutraStar Inc. and sold by CuraLife; it is a blend of nine ayurvedic plants and herbs.
  The CuraLin formulation contains the following ingredients (per 2 capsules):
  * Mormordica charantia (fruit) - 300mg
  * Gymnema sylvestre (leaf) - 80mg
  * Trigonella foenum-Graecum (seed) - 100mg
  * Curcuma longa (rhizome) - 100mg
  * Phyllanthus embilica officinalis (fruit) - 100mg
  * Swertia chiraytia (leaf) - 80mg
  * Syzgium Cumini (seed) - 100mg
  * Neopicrorhiza Picrorhiza/Scrophulariiflora Kurroa (root) - 100mg
  * Cinnamoum verum/zeylanicum - 40 mg
  * Hydroxypropyl methylcellulose
  * Rice Flour

SUMMARY:
The purpose of this study is to provide preliminary data necessary for a larger, controlled trial of CuraLin as a treatment option for T2DM. This study will also fill the gap in literature surrounding herbal medicine in the treatment of T2DM. The use of herbal preparations for diabetes has increased globally, and given the costs, adverse effects, lack of clinical outcome improvement, and minimal A1c reductions associated with medications, safer, more affordable alternatives need to be explored. CuraLin™ is a dietary supplement manufactured by NutraStar Inc. and sold by CuraLife; it is a blend of nine ayurvedic plants and herbs taken three times daily, after meals for the management of diabetes. It is hypothesized that CuraLin will be safely tolerated among adults with Type 2 Diabetes Mellitus, and will improve glucose control and cardiometabolic risk factors over this 12 week study.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults ≥18 and ≤ 75 years of age.
* Have an existing diagnosis of type 2 diabetes without known complications; i.e. eye damage (retinopathy), nerve damage (diabetic peripheral neuropathy), kidney damage (diabetic kidney disease), or heart damage (recent myocardial infarction or severe congestive heart failure).
* Must be on a stable dose (i.e. consistent dose for three months or greater) of all medications.
* Must be on a stable dose of dietary supplements for one month prior to enrollment.
* Have a serum hemoglobin A1c between 7% and 9.5%.
* Able to communicate via email, fill out a computer-administered questionnaire, and to read and write in English.
* Willing to have blood drawn at 3 separate time points.
* Willing to take an herbal supplement three times a day, daily, for 12 weeks.
* Willing to abstain from new anti-diabetic therapies, vitamins, minerals, dietary supplements, and lipid-lowering agents for 12 weeks.
* Willing and able to follow the study protocol and attend study visits.
* Approved to be eligible for study participation at the discretion of the Principal Investigators, after review of the Formal Eligibility Screen results.

Exclusion Criteria:

* Allergy to any ingredient found in the study product (Mormordica charantia (fruit), Gymnema sylvestre (leaf), Trigonella foenum-Graecum (seed), Curcuma longa (rhizome), Phyllanthus embilica officinalis (fruit), Swertia chiraytia (leaf), Syzgium Cumini (seed), Neopicrorhiza Picrorhiza/Scrophulariiflora Kurroa (root), Cinnamoum verum/zeylanicum, Hydroxypropyl methylcellulose, Rice Flour).
* Current use of insulin.
* Current use of CuraLin or any dietary supplement that has the same ingredients as CuraLin (see list of ingredients above).
* Current use of the following lipid-lowering medications: Ezetimibe (Zetia), Cholestyramine (Prevalite, Questran, Questran Light), Colesevelam (Welchol), or Colestipol (Colestid, Colestid Flavored).
* History of myocardial infarction or stroke within the last 6 months, current coronary artery disease, unstable angina, uncontrolled hypertension (i.e. systolic > 180 or diastolic > 110), congestive heart failure, or stated history of coronary bypass surgery or heart stent placement.
* Current active diabetic ulcers or history of diabetic neuropathy.
* Active malignancy, with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix.
* Current diagnosis of Small Intestinal Bacterial Overgrowth (SIBO), Small Intestinal Fungal Overgrowth (SIFO), Inflammatory Bowel Disease (IBD; i.e. Crohn's or Ulcerative Colitis), or other diagnosed pathology of the gastrointestinal tract (excluding Irritable Bowel Syndrome, [IBS]).
* Presence of an unstable and/or significant medical disorder that would compromise the participant's safety to take part in the study.
* Planned elective surgery within the next 12 weeks.
* Pregnant, nursing, or planning a pregnancy within the next 12 weeks.
* Women of childbearing age not using standard birth control measures.
* History of liver and/or kidney disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | 12 Weeks
  Hemoglobin is the oxygen-carrying component of red blood cells. In the presence of sustained elevated glucose levels, glucose non-enzymatically binds to hemoglobin, leading to the formation of glycated hemoglobin, and later, advanced glycation end products (AGEs). AGEs are responsible for many of the complications of T2DM. Thus, HbA1c, in conjunction with fasting blood glucose, is used as diagnostic criteria for T2DM (HbA1c ≥ 6.5%), and is used as a marker of glycemic control in diabetic individuals. As the life cycle of a red blood cell is approximately 90 days, serum HbA1c measurements are a snapshot of the percent of glycated hemoglobin over the prior two to three months, and thus serve as a snapshot of glycemic control in T2DM. HbA1c will be expressed as a percentage.
Gamma-glutamyltransferase (GGT) | 12 Weeks
  Concentration of the enzyme Gamma-glutamyltransferase (GGT) in the blood is considered a measure of liver inflammation and oxidative stress. Liver function markers will be expressed as IU/L.
Aspartate aminotransferase (AST) | 12 Weeks
  Concentration of the enzyme aspartate aminotransferase (AST) in the blood is considered a measure of liver inflammation. Liver function markers will be expressed as IU/L.
Alanine aminotransferase (ALT) | 12 Weeks
  Concentration of the enzyme alanine aminotransferase (ALT) in the blood is considered a measure of liver inflammation. Liver function markers will be expressed as IU/L.
Homeostatic Model Assessment of Insulin Resistance | 12 Weeks
  The Homeostatic model assessment (HOMA) of β- cell function and insulin resistance (IR) is a calculated ratio of fasting plasma insulin to glucose, and reflects the balance between hepatic glucose output and β- cell insulin secretion. It has been used in greater than 500 research publications to provide an estimate of insulin sensitivity and β- cell function, and is used to predict the level of insulin resistance. In patients with T2DM, the HOMA-IR is able to assess changes in β-cell function and IR, and thus, provide a reflection of treatment effects. The HOMA-IR will be expressed as a number, where '1' is considered normal, and anything above '1' is reflective of some degree of insulin resistance.

SECONDARY OUTCOMES:
Fasting Blood Glucose | 12 Weeks
  FBG, in conjunction with HbA1c, is used as a diagnostic criteria for T2DM (FBG ≥ 126 mg/dL), and is used as a marker of glycemic control in diabetic individuals. Levels are associated with future cardiac events and other complications of T2DM. FBG will be expressed in mg/dL.
Estimated glomerular filtration rate | 12 Weeks
  As estimation of the rate at which the kidneys filter and reabsorb protein based on age, ethnicity and blood creatinine.
Triglycerides | 12 Weeks
  The concentration of triglyceride-based fats in the blood is a cardiovascular risk factor.
LDL:HDL ratio | 12 Weeks
  The ratio of the concentration of low density lipoproteins (LDL) to high density lipoproteins (HDL) is a cardiovascular risk factor.
BMI | 12 Weeks
  Elevated body weight, manifesting as being overweight or obese, can cause and/or lead to exacerbations in a variety of pathologies, including T2DM, dyslipidemia, liver dysfunction, renal dysfunction, and cardiovascular disease. Thus, changes in weight are clinically meaningful in a T2DM population. This outcome measure is an important correlate and is of low burden to participants. Additionally, we will measure height in order to calculate Body Mass Index (BMI). Body weight will be expressed in pounds, height in inches, and BMI in kg/m2.
Creatinine | 12 weeks
  The concentration of creatinine in the blood is a measure of renal function.
Blood urea nitrogen (BUN) | 12 weeks
  The concentration of urea-based nitrogen in the blood is a measure of renal function.

OTHER OUTCOMES:
PROMIS-29 Health-related Quality of Life | 12 Weeks
  PROMIS-29 will measure health-related quality of life and is a validated, 29 question survey divided into seven sub-domains of function including physical functioning, social function, pain interference, pain intensity, sleep, depression, and anxiety.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National University of Natural Medicine, Portland, Oregon
  - Institute of Complementary Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No